CLINICAL TRIAL: NCT05882422
Title: Evaluation of the Effect of Dietary Phytochemical Index and Antioxidant Capacity on the Outcome of Ongoing Pregnancy in In Vitro Fertilization Treatment
Brief Title: Evaluation of the Effect of Dietary PI and TAC on the Outcome of Pregnancy in In Vitro Fertilization Treatment
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nagihan Kırcali Haznedar, Research Assisstant, Hacettepe University
Other Study IDs: 222S315
Record Dates: First submitted 2023-05-17; First posted 2023-05-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Ongoing Pregnancy; In-vitro Fertilization
Keywords: Phytochemicals; Polyphenols; Dietary İnflammatory Index; In-vitro fertilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to determine the relationship between dietary total antioxidant capacity, phytochemical index, inflammatory index, dietary polyphenol intake and ongoing pregnancy outcome in couples receiving IVF treatment.

In this context, the objectives are:

Determining the relationship between diet's antioxidant capacity, phytochemical index, inflammatory index, and dietary polyphenol intake and ongoing pregnancy outcome, Determining the relationship between total serum antioxidant capacity, serum oxidant capacity and CRP levels and ongoing pregnancy outcome, It is the determination of the relationship between body composition and ongoing pregnancy.

With this study, it is aimed to obtain reliable data on the effects of diet's antioxidant capacity, phytochemical index and dietary polyphenol intake and inflammatory index on reproductive functions. In this way, it is thought that nutritional recommendations that can be given to patients who will undergo IVF treatment before treatment will be developed.

In this study, which is a first in terms of examining many parameters related to diets of women and men, it will be evaluated whether the parameters to be examined are effective in IVF cycles.

The aims, objectives and hypotheses the researchers put forward within the scope of the study have not been studied extensively before. If the planned project is carried out successfully, new nutritional approaches will be paved in in-vitro fertilization treatment, and it will be possible to contribute to reducing the financial burden of the treatment. In addition, an important step will be taken to increase the total fertility rate (number of children per woman) within the scope of the 11th Development Plan (2019-2023). It also conforms to the 3rd Sustainable Development Goals, "healthy and quality life" (UNDP Turkey 2018)

ELIGIBILITY:
Inclusion Criteria:

* Females <41 years
* Males < 55 years
* BKI ≤ 32 kg/m2

Exclusion Criteria:

* Smoking cigarettes
* Chronic and inflammatory diseases
* Dietary changes in last 6 months
* Using antioxidant supplements
* Females diagnosed with infertility for anatomical reasons, endometriosis, tubal factor, or low ovarian reserve
* Males diagnosed with azospermia
* Couples who have had more than two failed cycles

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Couples who apply to the IVF unit and meet the following criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 1 year
  "Ongoing pregnancy" is a term used in reproductive medicine to describe a pregnancy that has progressed beyond the early stages and is continuing to develop with a viable fetal heartbeat. Ongoing pregnancy is typically confirmed by ultrasound examination after the gestational age of 12 weeks. In assisted reproductive technology (ART) cycles, ongoing pregnancy rate is an important outcome measure used to assess the success of the procedure, as it reflects the number of pregnancies that have the potential to result in live births.

SECONDARY OUTCOMES:
Clinical pregnancy | 1 year
  "Clinical pregnancy" is a term used in reproductive medicine to describe a pregnancy in which there is evidence of a gestational sac or fetal heartbeat on ultrasound examination. Clinical pregnancy is typically confirmed around 6-7 weeks of gestation and is a significant milestone in assisted reproductive technology (ART) cycles. The clinical pregnancy rate is often used as an outcome measure to assess the success of ART procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe, Ankara, Altındag, Turkey (Türkiye)